CLINICAL TRIAL: NCT06418594
Title: Adebrelimab Plus Apatinib and Etoposide for the Treatment of HER2-Negative Breast Cancer Brain Metastasis: A Phase II Study
Brief Title: Adebrelimab Plus Apatinib and Etoposide for the Treatment of HER2-Negative Breast Cancer Brain Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Wang Tao, Professor, Beijing 302 Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-070
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: HER2-negative Breast Cancer Brain Metastases
MeSH Terms: interventions — apatinib; Etoposide

STUDY DESIGN:
Intervention Model Description: This study adopts a single-arm, open-label design, planning to enroll 30 patients with HER2-negative breast cancer brain metastasis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab+Apatinib+Etoposide (Experimental): Adebrelimab: 1200mg， ivgtt，administered on the first day of each cycle, with a cycle of 21 days.
  Apatinib: 250 mg, oral, once daily, continuous use, with a cycle of 21 days.
  Etoposide: 50mg/day, oral, administered on days 1-14 of each cycle, with a cycle of 21 days.
  Interventions: Drug: Adebrelimab; Drug: Apatinib; Drug: Etoposide

INTERVENTIONS:
Drug: Adebrelimab — Adebrelimab: 1200mg, ivgtt, administered on the first day of each cycle, with a cycle of 21 days
Drug: Apatinib — Apatinib: 250 mg, oral, once daily, continuous use, with a cycle of 21 days
  Other Names: Apatinib Mesylate Tablets
Drug: Etoposide — Etoposide: 50mg/day, oral, administered on days 1-14 of each cycle, with a cycle of 21 days
  Other Names: VP-16

SUMMARY:
Some studies have shown that approximately 15% of patients with advanced hormone receptor (HR) positive breast cancer and 1/3 of triple negative breast cancer will develop brain metastasis. At present, there is no unified drug treatment standard for HER2-negative breast cancer brain metastasis (BCBM). The evidence of single traditional chemotherapy drug as the main treatment of brain metastasis is not sufficient. Some exploratory studies on HER2-negative BCBM have shown that the central nervous system objective response rate (CNS-ORR) of anti-angiogenic drugs combined with chemotherapy is around 55%-80%。 Adebrelimab (a humanized PD-L1 monoclonal antibody) specifically blocks the binding of PD-1 and PD-L1, terminates the immunosuppressive signal produced by T cells, and makes T cells re-recognize tumor cells and kill them, thereby inhibiting tumor growth. In China, Adebelizumab has been approved for using in combination with chemotherapy as a first-line treatment for extensive stage small cell lung cancer. Apatinib (a small molecule VEGFR tyrosine kinase inhibitor) mainly plays an anti-angiogenic effect in the treatment of malignant tumors by inhibiting VEGFR. Apatinib has been approved monotherapy for advanced gastric adenocarcinoma or gastroesophageal junction adenocarcinoma that has progressed or relapsed after at least two systematic chemotherapies, advanced liver cancer that has failed or is intolerable after at least first-line systematic treatment, and first-line treatment in patients with unresectable or metastatic hepatocellular carcinoma combined with camrelizumab.

Due to the lack of effective drug therapy for HER2-negative BCBM, a variety of treatment combinations are still being explored. We hypothesized that adebrelimab plus apatinib and etoposide is an explorable and effective treatment for HER2- negative BCBM.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥18 years
* Expected survival time ≥3 months.
* Histologically or cytologically confirmed HER2-negative (IHC 0 or 1+; or IHC 2+ ISH negative) locally recurrent or metastatic disease
* New brain metastasis or brain metastasis progression after treatment
* HR+ advanced breast cancer with prior CDK4/6 inhibitor treatment failure or the investigator deems unsuitable for CDK4/6 inhibitors
* At least one intracranial measurable lesion as defined by RECIST V1.1 criteria；
* ECOG PS 0-2；
* Patients must have the ability to swallow oral medication；
* Prior WBRT, stereotactic radiosurgery, and surgical resection are allowed；
* Organ function levels are basically normal, and the investigator believes that the study drug can be applied：
* Voluntarily join this study, sign the informed consent, have good compliance, and are willing to cooperate with follow-up

Exclusion Criteria:

* Urgent need for local treatment of brain metastasis
* Immunohistochemistry HER2 positive (IHC 3 or IHC 2 ISH amplification)
* Previously treated with Apatinib, Avelumab, or VP-16；
* Severe dysfunction of important organs such as the heart, liver, or kidneys；
* Inability to swallow, chronic diarrhea, and intestinal obstruction, with multiple factors affecting drug administration and absorption；
* Participants diagnosed with any other malignant tumor within 5 years before this study, excluding non-melanoma skin cancer that has undergone radical treatment. Basal cell or squamous cell skin cancer or cervical carcinoma in situ and thyroid papillary carcinoma。
* Patients who allergy to any component of the drugs in this protocol; patients with history of immunodeficiency, including HIV positive, HCV, active hepatitis B, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation
* History of any cardiac disease, including: (1) arrhythmia requiring medication or clinically significant; (2) myocardial infarction; (3) heart failure; (4) any other cardiac disease judged by the investigator to be unsuitable for participation in this trial, etc.
* Pregnant or lactation female patients; females of childbearing age with a positive baseline pregnancy test or unwilling to take effective contraceptive measures during the entire trial period；
* According to the investigator's judgment, there are severe accompanying diseases that endanger the patient's safety or affect the completion of the study (including but not limited to uncontrolled severe hypertension, severe diabetes, active infection, etc.).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CNS-ORR | 2 months
  Central nervous system objective response rate (CNS-ORR), as assessed according to the RANO-BM criteria

SECONDARY OUTCOMES:
CNS-PFS | 1 Year
  CNS progression-free survival
Extracranial objective response rate | 2 Years
  According to recist1.1 standard, the proportion of patients whose extracranial best remission was CR or PR accounted for the total number of evaluable patients
Extracranial progression-free survival | 2 Years
  The time to the date of first documented progression or date of death from any cause, whichever came first
OS | 3 Years
  The time from the beginning of treatment to the time of death caused by any cause
CBR | 2 Years
  Clinical benefit rate: CR+PR+SD≥6 months
DoR | 2 Years
  The time from the beginning of CR or PR to the time when the tumor was first evaluated as PD or any cause of death.
Safety | AE recorded from infromed consent to 28 days after treatment completion
  Adverse events (AE), serious adverse events (SAE), and immune-related adverse events (irAE), in accordance with the NCI-CTC AE version 5.0 criteria. AE recorded from infromed consent to 28 days after treatment completion.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China